CLINICAL TRIAL: NCT05976360
Title: A Randomized, Open-label, Parallel Design Study of the Pharmacokinetics, Tolerability and Safety of Two Different Dupilumab Drug Products After Administration of Single Subcutaneous Doses
Brief Title: A Study to Investigate the Pharmacokinetics, Tolerability and Safety of Two Different Dupilumab Drug Products in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKM14161; U1111-1290-9436 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07-24

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Dupilumab drug product 1 (Active Comparator): A single subcutaneous injection on Day 1
  Interventions: Drug: Dupilumab (SAR231893)
- Dupilumab drug product 2 (Experimental): A single subcutaneous injection on Day 1
  Interventions: Drug: Dupilumab (SAR231893)

INTERVENTIONS:
Drug: Dupilumab (SAR231893) — Injection solution, subcutaneous
  Other Names: REGN668
  Arms: Dupilumab drug product 1
Drug: Dupilumab (SAR231893) — Injection solution, subcutaneous.
  Other Names: REGN668
  Arms: Dupilumab drug product 2

SUMMARY:
This is a phase 1, single subcutaneous dose study to evaluate safety and pharmacokinetics of 2 different dupilumab drug product in healthy volunteers. The duration per participant is up to 11 weeks.

DETAILED DESCRIPTION:
Duration per participant is up to 11 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, between 18 and 65 years of age, inclusive.
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
* Body weight between 70.0 and 90.0 kg, inclusive.
* Having given written informed consent prior to undertaking any study-related procedure.

Exclusion Criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease, or signs of acute illness.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month).
* Blood donation or collection totaling more than 250 mL (including collections during study screening) within 2 months before inclusion on Day -1.
* Symptomatic postural hypotension, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥20 mmHg within 3 minutes when changing from supine to standing position.
* History of light-headedness or syncope during blood collection or injection of medications.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.
* History or presence of drug or alcohol abuse (alcohol consumption more than 40 g per day on a regular basis).
* If female, pregnancy (defined as positive β-human chorionic gonadotropin blood test) or breast-feeding.
* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease, or signs of acute illness.
* Participation in any clinical research study evaluating another investigational drug or therapy within 30 days or 5 elimination half-lives of the respective investigational drug, whichever is longer, of the inclusion visit.
* Any participant who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-11-02 (Actual); Primary Completion 2015-01-17 (Actual); Study Completion 2015-01-17 (Actual)

PRIMARY OUTCOMES:
Maximum serum concentration observed: Cmax | Up to Day 57
Time to reach Cmax (tmax) | Up to Day 57
Area under the serum concentration versus time curve from time zero to the real time of last measurable concentration (AUClast) | Up to Day 57

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Up to Day 57
Incidence of anti-dupilumab antibodies (ADA) | Up to Day 57

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Prism Research-Site Number:840002, Saint Paul, Minnesota
  - Biokinetic Clinical Applications-Site Number:840003, Springfield, Missouri

IPD SHARING:
Plan to Share IPD: No